CLINICAL TRIAL: NCT06895187
Title: Catheter Ablation Using a Novel Navigation and Imaging System
Acronym: ENVIsIoN
Status: Not yet recruiting | Type: Observational
Sponsor: LUMA Vision Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ENVISION-P003
Record Dates: First submitted 2025-03-24; First posted 2025-03-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: VERAFEYE System — VERAFEYE system guidance will be used on all patients undergoing PAF ablation.

SUMMARY:
The objective of the ENVIsIoN study is to collect data on the use of the VERAFEYE navigation and imaging system in patients indicated to undergo a catheter ablation procedure for the treatment of Paroxysmal Atrial Fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age at the time of consent, or of legal age to give informed consent specific to state and national law
* Subjects is eligible for a catheter ablation procedure with the VERAFEYE System as navigation and imaging system in the treatment of PAF (according to VERAFEYE System IFUs, current international and local guidelines and per physician discretion)
* Subject is able to understand and willing to provide written informed consent
* Subject is able to and willing to complete all study assessments associated with this clinical study at an approved clinical investigational center

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Subjects who have undergone a previous cardiac ablation for the treatment of PAF
  * Subject where placement of VERAFEYE Imaging Catheter is technically not feasible per physician discretion
  * Pregnant women or women who plan to become pregnant during the course of their participation in the study (women should either be of non- childbearing potential at the time of enrolment (as documented in the medical file) or have a negative pregnancy test within the previous 7 days prior to the procedure)
  * Unrecovered/unresolved Adverse Events from any previous invasive procedure
  * Subjects who are currently enrolled in another study (except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Acute procedural success rates during the index procedure | During the procedure
  A procedure will be defined as successful if all the following conditions occur during the case:
  * ability to create a 3D anatomical model with the VERAFEYE System and
  * completion of the necessary ablation applications for PAF using the 3D anatomical model created with the VERAFEYE System

IPD SHARING:
Plan to Share IPD: No